CLINICAL TRIAL: NCT05545514
Title: Individualized Homeopathy to Reduce the Use of Antibiotics in Women With Recurrent Uncomplicated Urinary Tract Infections
Acronym: iHOM
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: School of Medicine, Technical University Munich, Münchner Studienzentrum (Unknown); Klinikum rechts der Isar, TUM Institute for AI and Informatics in Medicine (AIIM) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IHO-0000-REN-0220-S
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-04

CONDITIONS: Urinary Tract Infection Chronic
Keywords: Cystitis; Nephritis
MeSH Terms: conditions — Cystitis; Nephritis | interventions — Taste

STUDY DESIGN:
Intervention Model Description: Phase IV, monocentric, randomised, double-blind, parallel-group, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Individualized homeopathy (iHOM):
  One out of 140 predefined homeopathic medical products (HMP) in potency C200 or C1000, individually selected as indicated per homeopathic treatment principles. The HMPs are sucrose pillules, impregnated with the specific homeopathic substance and potency and will be administered once at baseline: 5 pillules sublingually. The dosage of the HMP can be repeated or adapted according to the homeopathic treatment principles three times during the course of the study and, in addition, in the event of an acute UTI.
  Interventions: Drug: One out of 140 predefined homeopathic medical products (HMP) in potency C200 or C1000,
- Placebo (Placebo Comparator): Non-impregnated sucrose pillules, identical to the HMP (verum) in appearance, taste and size.
  Interventions: Drug: One out of 140 predefined homeopathic medical products (HMP) in potency C200 or C1000,

INTERVENTIONS:
Drug: One out of 140 predefined homeopathic medical products (HMP) in potency C200 or C1000, — To investigate the efficacy of individualised homeopathic treatment (potency C200 and/or C1000) in comparison to placebo regarding the number of UTI treated with antibiotic agents.
  Other Names: Placebo; Non-impregnated sucrose pillules, identical to the HMP (verum) in appearance, taste and size.

SUMMARY:
The aim of the study is to determine the efficacy of individualised homeopathic drug treatment (potency C200 and C1000) compared to placebo in females (age 18<65) with recurrent urinary tract infections, per definition ≥ 2 UTI in 6 months and/ or ≥ 3 UTI in 9 months.

DETAILED DESCRIPTION:
The World Health Organization has declared the problem of antibiotic resistance to be a global crisis and the European Union has defined, among other things, the reduction of antibiotic use in its strategies to avoid the development of resistance. Recurrent UTIs are one of the most common infectious diseases contributing to a multiple of multidrug- resistant extra intestinal pathogenic E coli, increasing morbidity and mortality due to many treatment failures and hospital admissions, which leads to increased healthcare costs. There is, therefore, an urgent need to optimize appropriate usage, in order to minimize the burden of disease for the patients and the health care services, while maintaining treatment safety at the same time.

In Germany, it is currently recommended to treat uncomplicated UTIs symptomatically as long as no dangerous course of the disease can be expected, but different treatment options aiming to decrease the frequency of UTI treated with antibiotics have shown only limited success. Thus, the symptom load of the affected patients as well as prescription rates for antibiotics remain high and treatment options are warranted by patients and physicians.

Homeopathy has shown relevant clinical effects for other recurrent infectious diseases and a reduction of the frequency of recurrent UTIs with individualised homeopathic treatment (iHOM) has been observed in practice. In this study we therefore aim to test the efficacy of this treatment approach as an add-on therapy to the treatment standard in a double-blind, placebo-controlled randomised clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Females, age 18 < 64 years
2. Signed informed consent
3. Documented recurrent UTI (i.e. ≥ 2 UTI in 6 months and/ or ≥ 3 UTI in 12 months)
4. No change of other prophylactic treatment (e.g. Urovaxom, oestrogen) for recurrent UTI for at least three months before baseline
5. No product or dosage change of systemic hormonal treatment (including oral anticonception) for at least three months before baseline
6. Female participants who are not capable of bearing children or who use a method of contraception that is medically approved by the health authority of the respective country.

This includes:

* A woman who is not capable of bearing a child is defined as follows: post-menopausal (12 months natural (spontaneous) amenorrhea or 6 months spontaneous amenorrhea with serum-FSH-values (follicle-stimulating hormone) of >40 mIU/mL); 6 weeks after a bilateral ovariectomy with or without hysterectomy or sterilization by means of tubal ligation
* A woman capable of bearing child is defined as follows: a woman who is physiologically capable of becoming pregnant, including women whose occupation, lifestyle or sexual orientation exclude sexual intercourse with a male partner and women whose partners have been sterilized by vasectomy or other measures.
* Medically-approved methods of contraception can include the following: hormonal contraceptives, intrauterine device and double barrier method. Acceptable preventive measures can include total abstinence at the discretion of the investigator, in cases where compliance is ensured because of the study participant's age, occupation, lifestyle or sexual orientation. Periodical abstinence (e.g. calendar, ovulation, symptothermal methods or abstinence until the 4th day after the ovulation) as well as coitus interruptus are not acceptable methods of contraception.
* A reliable method of contraception must be used for the entire duration of the study.

Exclusion Criteria:

1. Individual symptomatology of the patient indicates the prescription of a HMP which is not available within this clinical trial 2. Pregnancy or breast feeding after pregnancy 3. Women with a complicated urinary tract infection (including infections occurring due to anatomical abnormalities (e.g. an obstruction, renal tract calculi, hydro nephrosis), infections occurring due to an immune compromised state (e.g. HIV, immune suppressive therapy), and recurrent infections despite adequate treatment (multi-drug resistant organisms or atypical organisms)) 4. Surgery of the urinary tract or the pelvic floor 5. Known hypersensivity against the study medication or the recommended on demand medication (Ibuprofen) 6. Homoeopathic therapy for recurrent UTIs during the last 6 months before baseline 7. Postmenopausal woman WITHOUT previous attempt of a therapy with locally applicate (vaginal) oestrogen 8. Serious acute or chronic organic disease or serious mental disorder, including

* diseases requiring immune suppressive therapy
* diabetes mellitus type 1 or 2 with an HbA1c > 7%
* any acute organic failure
* any advanced chronic organic failure (e.g. grade 3 or more)
* active cancer
* active (=clinically unstable) epileptic, cardiovascular or other organic pathology 9. Patients not able to declare meaningful informed consent on their own (e.g. with legal guardian), or other vulnerable patients (e.g. under arrest) 10. Simultaneous participation in any other clinical trial 11. Employees or family members of the sponsor or investigators

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
ICIQ-FLUTS: | Baseline to month 9
  To compare the number of UTI treated with antibiotic agents, measured between Baseline and month 9 in both groups
  A UTI is defined by the criteria of the German S3-guideline for the diagnostic of uncomplicated lower UTI:
  1. Clinical symptoms (either dysuria or increased urinary frequency or increased incontinence or pelvic pain) plus > 103 bacteria as monoculture in the urine culture, or
  2. Clinical symptoms plus urine test-strip with an evidence of nitrite and / or leukocyte-esterase and/ or blood
  The criteria for a prescription of antibiotic agents to the patient are:
  1. Fever > 38.0 degree Celsius, and / or
  2. Persistent pain under symptomatic therapy with Ibuprofen, not tolerated by the patient, and / or
  3. Clinical suspicion of pyelonephritis

SECONDARY OUTCOMES:
ICIQ-FLUTS and ACSS | Baseline to 6 month
  Time until the first UTI after the start of the study treatment (regardless of treatment of the first UTI)
ICIQ-FLUTS and ACSS | measured between Baseline and month 9
  The number of UTI treated with antibiotic agents
ICIQ-FLUTS and ACCS | measured between Baseline and month 9
  The number of UTI treated symptomatically
SF 12 | measured at Baseline and month 9 per visual analogue scale (VAS)
  Subjective symptom load and disease-specific quality of life over the last 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Renders, Prof. Dr. med., Principal Investigator — Klinikum rechts der Isar, TUM, Department Nephrology
Locations (1):
- Klinikum rechts der Isar, Department of Nephrology, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No